CLINICAL TRIAL: NCT02193906
Title: Neuropsychological Profile of a Portuguese Patient's Group With Multiple Sclerosis and Results of a Cognitive Rehabilitation Program
Brief Title: Neuropsychological Profile of a Patient's Group With Multiple Sclerosis and Effect of a Cognitive Rehabilitation Program
Acronym: MS_Rehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Ivânia A Alves, MD, MD, Campus Universitário de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSR-2013
Record Dates: First submitted 2013-09-18; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Cognitive Dysfunction
Keywords: Cognitive training; Multiple sclerosis; Cognitive deficits
MeSH Terms: conditions — Cognitive Dysfunction; Multiple Sclerosis; Cognition Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Cognitive training.
  Interventions: Other: Cognitive training
- Placebo group (Placebo Comparator): Placebo task.
  Interventions: Other: Placebo task

INTERVENTIONS:
Other: Cognitive training — Every patient will have 3 neuropsychological evaluations (with the same battery): baseline, after a 3-month period of training and 6 months after the conclusion of the training. Patients who have computer with internet access at home will perform a minimum of 3 sessions per week of Cogweb® during 3 months. Patients who don't have computer with internet access at home will perform a minimum of 3 sessions per week of Cogweb Monthly Notebooks® during 3 months. Every patient included will have an outpatient appointment in the end of the first and second months of training.
  Arms: Intervention group
Other: Placebo task — Every patient will have 3 neuropsychological evaluations (with the same battery): baseline, after a 3-month period of training and 6 months after the conclusion of the training. Patients will have to complete a placebo task (send an email with a copy of a journal/magazine heading) a minimum of 3 times a week, for 3 months. Every patient included will have an outpatient appointment in the end of the first and second months of training.
  Arms: Placebo group

SUMMARY:
The purpose of the study is to determine the effect of an web-based intensive cognitive rehabilitation program in neuropsychological performance of a population of patients with multiple sclerosis or clinical isolated syndrome.

DETAILED DESCRIPTION:
Objectives

Primary:

1. To determine the effect of an intensive cognitive rehabilitation program in neuropsychological performance of a population of patients with multiple sclerosis or clinical isolated syndrome.

Secondary:

1. To characterize the neuropsychological profile of a population of patients with multiple sclerosis or clinical isolated syndrome.
2. To evaluate the relation between Expended Disability Status Scale score and cognitive dysfunction.
3. To evaluate the impact of depression on neuropsychological performance.
4. To evaluate the relation between cognitive dysfunction and the 9-hole peg test.
5. To evaluate the relation between cognitive dysfunction and the 25-foot walk test.

Population and Sample Patients will be selected from an electronic database that exists in Centro Hospitalar Entre Douro e Vouga. They will be consecutively convoked and it will be proposed neuropsychological evaluation and participation in the study.

Every patient will have a baseline neuropsychological evaluation (table 1). After that, they will be randomized for training (Cogweb® program or Cogweb Monthly Notebooks®) or placebo in a 2(training):1(placebo) fashion (online program of randomization). After a 3-month period of tasks (training versus placebo), they will have another neuropsychological evaluation with the same battery used for baseline.

Patients included in intervention arm that have computer with internet access at home will perform a minimum of 3 sessions per week of Cogweb® during 3 months. Patients included in intervention arm that don't have computer with internet access at home will perform a minimum of 3 sessions per week of Cogweb Monthly Notebooks® during 3 months.

Patients included in placebo arm will have to complete a task (send an email with a copy of a journal/magazine heading) a minimum of 3 times a week.

Every patient included will have an outpatient appointment in the end of the first and second months of tasks (training versus placebo).

The placebo group is a group of patients with multiple sclerosis, selected according to inclusion and exclusion criteria, from the same database than those assigned for training.

The neuropsychological evaluation plan comprises: global efficiency (Montreal Cognitive Assessment test); processing speed (reading task of Stroop test, symbol searching from Wechsler Adult Intelligence Scale); attention (letter cut of Behavioural Inattention Test, Trail making test part B); memory (Letter and number sequence of Wechsler Memory Scale, digit memory, spatial localization of Wechsler Memory Scale, logic memory of Wechsler Memory Scale, word list from Wechsler Memory Scale); executive functions (colour naming task of Stroop test, inhibition from INECO frontal screening, verbal initiative from Lisbon Dementia Evaluating Battery, Zoo Map from Ineco, Matrix from Wechsler Adult Intelligence Scale) and anxious and depressive symptoms (Hospital Anxiety and Depression Scale).

Sample Size There will be convoked 75 patients (convenience sample).

Design Experimental, single-center study.

Clinical Practice Concomitant medication allowed Any except corticotherapy. Discontinuation criteria

1. Desire of the patient to end participation in the study.
2. Noncompliance of the intervention plan or fail the appointments predetermined.

Parameters to evaluate de study objectives

1. Neuropsychological battery: performed at baseline and at 3 months after the completion of study tasks (each test is composed of numerical, continuous variables).
2. Expended Disability Status Scale score: screening at baseline.
3. Stage of the disease: screening from the database.
4. Number of years of disease evolution.
5. 9-hole peg test: performed at baseline and at 3 months after the completion of study tasks.
6. 25-foot walk test: performed at baseline and at 3 months after the completion of study tasks.

Efficacy Endpoints Primary: To determine if an intensive cognitive rehabilitation program changes, in a statistically significant way, the performance on a neuropsychological evaluation after 3 months of training, comparing to the control group (number of tests scored more than one standard deviation from the normal value). There will be analyzed the total and partial scores for each test. The individuals with cognitive deficits at baseline will be analyzes as rehabilitation group. The others (without cognitive deficits in cognitive evaluation at baseline) will be analyzed as a separated group of cognitive stimulation.

Secondary:

1. To characterize the profile of a population of patients with multiple sclerosis, according to the performance in a neuropsychological battery, in terms of processing speed, attention, memory and executive functions.
2. To determine the percentage of patients with Cognitive Dysfunction, defined as performance >1standard deviation below the median in ≥3 tests of the battery.
3. To correlate the Expended Disability Status Scale score with the Cognitive Dysfunction.
4. To correlate the Hospital Anxiety and Depression Scale score with the Cognitive Dysfunction.
5. To correlate the 9-hole peg test with the Cognitive Dysfunction.
6. To correlate the 25-foot walk test with the Cognitive Dysfunction.

Safety Endpoints Not applicable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MS diagnosed according to McDonald criteria from 2010 and clinical isolated syndrome patients.
* Age ≥18 years old.
* Informed consent.

Exclusion Criteria:

* Disease relapse in the last month.
* Corticotherapy in the last month.
* Expended Disability Status Scale score >6,0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Effect of an intensive cognitive rehabilitation program in neuropsychological performance of a population of patients with multiple sclerosis or clinical isolated syndrome. | 3 months
  Two neuropsychological assessments were made: at baseline and at 3 months with the same neuropsychological battery to all the patients.
  After that, the statistically significant differences between the two study groups (comparing the standard deviations from the normative values of each test), will be accessed. The tests will be analysed separately and globally as a battery.

SECONDARY OUTCOMES:
Neuropsychological profile of a population of patients with multiple sclerosis or clinical isolated syndrome. | Baseline
  Characterization of the cognitive profile of deficits in the following domains (percentage of deficits by domain, considering all patients who have done the baseline evaluation): global efficiency, processing speed, attention, memory and executive functions.
Percentage of patients with Cognitive Dysfunction | Baseline
  Patients with performance >1standard deviation below the median in ≥3 tests of the battery of neuropsychological evaluation will be considered as having Cognitive Dysfunction.
Relation between Expended Disability Status Scale score and cognitive dysfunction. | Baseline
  Patients with performance >1standard deviation below the median in ≥3 tests of the battery of neuropsychological evaluation will be considered as having Cognitive Dysfunction.
  Correlation between Expended Disability Status Scale score and Cognitive Dysfunction.
Impact of depression on neuropsychological performance. | Baseline
  Patients with performance >1standard deviation below the median in ≥3 tests of the battery of neuropsychological evaluation will be considered as having Cognitive Dysfunction.
  Correlation between Hospital Anxiety and Depression Scale score and Cognitive Dysfunction.
Relation between cognitive dysfunction and the 9-hole peg test. | Baseline
  Patients with performance >1standard deviation below the median in ≥3 tests of the battery of neuropsychological evaluation will be considered as having Cognitive Dysfunction.
  Correlation between 9-hole peg test time frame (in seconds) and Cognitive Dysfunction.
Relation between cognitive dysfunction and the 25-foot walk test. | Baseline
  Patients with performance >1standard deviation below the median in ≥3 tests of the battery of neuropsychological evaluation will be considered as having Cognitive Dysfunction.
  Correlation between 25-foot walk test time frame (in seconds) and Cognitive Dysfunction.

OTHER OUTCOMES:
Long term effects of an intensive cognitive rehabilitation program in neuropsychological performance of a population of patients with Expended Disability Status Scale. | 9 months
  Two neuropsychological assessments were made: at baseline and at 9 months with the same neuropsychological battery to all the patients included who performed the 3months cognitive training or placebo tasks.
  After that, the statistically significant differences between the two study groups (comparing the standard deviations from the normative values of each test), will be accessed. The tests will be analysed separately and globally as a battery.

CONTACTS AND LOCATIONS:
Overall Officials: Vitor T Cruz, MD, Study Director — Clinical Research Office - Health Sciences Department; Ivânia A Alves, MD, Principal Investigator — Clinical Research Office, Health Sciences Department